CLINICAL TRIAL: NCT03856749
Title: Effectiveness of Wheelchair Skills Training for Caregivers of Manual Wheelchair Users: a Randomized Waitlist-controlled Trial
Brief Title: Effectiveness of Wheelchair Skills Training for Caregivers of Manual Wheelchair Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lee Kirby (Other)
Collaborators: IWK Health Centre (Other)
Responsible Party: Sponsor-Investigator, Lee Kirby, Principal Investigator, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WSP2019-01
Record Dates: First submitted 2019-02-22; First posted 2019-02-27 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Caregivers

STUDY DESIGN:
Intervention Model Description: A single-blind randomized controlled trial. Each participant in the study consists of a caregiver and wheelchair user dyad. 1 dyad = 1 manual wheelchair user + his/her caregiver.
Who Masked: Outcomes Assessor
Masking Description: This is a single-blind study. The outcomes assessor will be blind to group allocation. Because of the nature of the study, it will not be possible to blind participants or trainer.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): The wheelchair user and caregiver will be trained together on wheelchair skills using remote technology (Zoom for healthcare and/or Facetime).
  Interventions: Other: Remote wheelchair skills training
- Control (No Intervention): The wheelchair user and caregiver will receive the same self-study materials provided to the Treatment arm. Usual care, which may include wheelchair skills training for both wheelchair users and caregivers( but which often does not do so to an adequate extent) by wheelchair user's clinical therapist.

INTERVENTIONS:
Other: Remote wheelchair skills training — Prior to the first training session, the trainer will be provided with the results from the assessment immediately preceding training to provide him/her time to individualize the training session. Trainer will provide self-study materials (the Caregiver Handbook and caregiver-training video-recording) and an explanation on how these materials should be used.
  The wheelchair user and caregiver will be trained together on wheelchair skills, using the principles of the Wheelchair Skills Training Program, as outlined in the Wheelchair Skills Program Manual using remote technology. Each training session will be with a trainer-to-dyad ratio of 1:1 1 dyad = 1 manual wheelchair user + his/her caregiver. Training will continue until the goals have been met and retained (for at least one subsequent session), using up to 4 training sessions that will each last up to 60 minutes at intervals a minimum of 3 days.
  Arms: Treatment

SUMMARY:
Although there have been a small number of studies suggesting the important role that caregivers play in assisting wheelchair users with mobility, there has never been a randomized controlled trial (RCT) looking at the effectiveness or cost-utility of wheelchair skills training for caregivers. The overall goal of this study is to correct this knowledge gap and, triggered by the COVID-19 pandemic of 2020, to conduct the training remotely. The main purpose of this study is to test if providing wheelchair skills training remotely to caregivers of manual wheelchair users enhances caregiver-assisted wheelchair skills ability and confidence in comparison to a control group of participants who are receiving usual care and self-study material on wheelchair skills. The investigators will also study whether the benefits of training are still seen at a 6-week follow-up and assess the health-economic impact of caregiver training.

ELIGIBILITY:
Inclusion Criteria for caregiver and wheelchair user dyad

* be ≥ 18 years of age
* able to communicate in English
* be willing to participate and be committed to setting regularly scheduled times for the study activities
* will need to have the appropriate connectivity for the remote training and testing (i.e. telephone, limited-access e-mail and internet).

Exclusion Criteria for caregiver and wheelchair user dyad :

* fail to complete the baseline (T1) assessment
* have unstable medical conditions (e.g. angina, seizures) that might make the use of a manual wheelchair dangerous
* emotional problems (e.g. severe anxiety, depression) that might make participation unsafe or unpleasant
* have a medical condition that is likely to deteriorate in the three months following enrollment.

Inclusion Criteria for wheelchair user

* a person who uses a manual wheelchair
* be expected to continue to use a manual wheelchair at least part-time in the coming months
* requires no more than minimal assistance for communication and auditory comprehension

Inclusion Criteria for caregiver of wheelchair user

-must be a caregiver (e.g. a family member, friend, volunteer or regular homecare worker) who spends an average total of at least 2 hours per week with the manual wheelchair user that includes manual wheelchair mobility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-12-04 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Wheelchair Skills Test Questionnaire at 5 weeks | 5 weeks
  Change from baseline in self-reported ability and confidence to perform 33 wheelchair skills. Score ranges from 0-100%, with 0 indicating a poor outcome (not able to do any wheelchair skills and 100% indicating being able to do all the skills).
Change from baseline in Wheelchair Skills Test Questionnaire at 18 weeks | 18 weeks
  Change from baseline in self-reported ability and confidence to perform 33 wheelchair skills. Score ranges from 0-100%, with 0 indicating a poor outcome (not able to do any wheelchair skills and 100% indicating being able to do all the skills).

SECONDARY OUTCOMES:
Satisfaction with wheelchair skills training over course of study | 5 weeks, 18 weeks
  Participants will be asked their perceptions of the content and benefits of the training material.
Cost-effectiveness of training | 5 weeks
  Measured using Quality-Adjusted Life Years (QALY), estimated costs and quality of life. QALY scores range from 0(dead) to 1(perfect health).
Change from baseline in quality of life at 5 weeks | 5 weeks
  Change from baseline in quality of life measured using the EQ-5D-5L as validated quality of life self-report outcome measure. Scores range from 1 (no problem) to 5 (extreme problem) in dimensions of mobility, self-care, activities, pain and mental health. General health score from 0 % (worst health imaginable) to 100% (best health imaginable).
Change from baseline in quality of life at 18 weeks | 18 weeks
  Change from baseline in quality of life measured using the EQ-5D-5L as validated quality of life self-report outcome measure. Scores range from 1 (no problem) to 5 (extreme problem) in dimensions of mobility, self-care, activities, pain and mental health. General health score from 0 % (worst health imaginable) to 100% (best health imaginable).

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Rehabilitation Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Kirby RL, Smith C, Miller MD, Osmond D, Sherman MA, Parker K, Koto PS, Theriault CJ, Sandila N. Wheelchair skills training for caregivers of manual wheelchair users: a randomized controlled trial comparing self-study and remote training. Disabil Rehabil Assist Technol. 2024 Nov;19(8):2896-2903. doi: 10.1080/17483107.2024.2321272. Epub 2024 Feb 29. PMID 38420947